CLINICAL TRIAL: NCT03361592
Title: Immediate Effects of Spinal Manipulative Therapy (SMT) on Kinetic and Kinematic Symmetry on Functional Performance Tests: a Test-retest, Single-blinded, Randomized Controlled Trial.
Brief Title: The Immediate Effects of Spinal Manipulative Therapy on Kinetic and Kinematic Symmetry.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Bruno Araújo Procópio de Alvarenga, PT, DC, Phd Student, Physiotherapist and Chiropractor, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ulisboa
Record Dates: First submitted 2017-11-06; First posted 2017-12-05 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Asymptomatic Condition
Keywords: symmetry index, functional performance tests, SMT
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Therapeutics; Manipulation, Spinal; salicylhydroxamic acid; Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled single-blinded study.
Who Masked: Outcomes Assessor
Masking Description: Participants were initially instructed about the study procedures with therapeutic interventions. After collected data, the participants were asked about the therapeutic intervention, if they are capable to identify which intervention were performed, SMT or SHAM, as parte of study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Manipulative Therapy (Experimental): The participants assigned to the intervention group received the procedure Lumbar (SMT) was performed after baseline measurements, using Diversified techniques, aiming to correct vertebral dysfunctional segments after clinical assessment. Participants were asked to lay down prone on, to perform spinal motion palpation analysis was performed in order to evaluate the presence of dysfunction in vertebral segments of lumbar spine.
  Interventions: Procedure: Spinal Manipulative Therapy
- Sham pre-load positioning SMT (Sham Comparator): The participants assigned to the control group received the procedure "Sham" (pre-load positioning MVT). The Sham (SMT) was performed with participant body positioning in the lateral position, as the SMT intervention. The doctor followed the participant through the same position of (SMT) intervention, using the maintenance of set-up position, but no manipulative thrust was delivered. The therapist applied minimal pressure and slid their hands across the skin to mimic the manipulative trust. The position was maintained for approximately 1 minute in total, 30 seconds on each side, and none of force or researcher body weight were putted in this procedure, only minimal pressure common to stabilize the set up position of (SMT).
  Interventions: Procedure: SHAM

INTERVENTIONS:
Procedure: Spinal Manipulative Therapy — Lumbar (SMT) was performed using Diversified techniques, aiming to correct vertebral dysfunctional lumbar segments. Participants were asked to lay down prone on, to perform spinal motion palpation analysis was in order to evaluate the presence of dysfunction in vertebral segments of lumbar spine.
  Other Names: Movement Disorders/therapy; Spinal Manipulation
  Arms: Spinal Manipulative Therapy
Procedure: SHAM — The "SHAM" (pre-load positioning SMT) was performed with participant body positioning in the lateral position, as the SMT intervention. The doctor followed the participant through the same position of (SMT) intervention, using the maintenance of set-up position, but no manipulative thrust was delivered. The therapist applied minimal pressure and slid their hands across the skin to mimic the manipulative trust. The position was maintained 30 seconds on each side, and none of force or researcher body weight were putted in this procedure, only minimal pressure common to stabilize the set up position of (SMT).
  Other Names: Control Group
  Arms: Sham pre-load positioning SMT

SUMMARY:
Athletes have been exposed to an ever increasing training load and subsequent biomechanical overload due to a constant demand for performance enhancement. As a result, it is observed an increased rate of musculoskeletal problems, including spinal biomechanical dysfunctions that are often asymptomatic. These dysfunctions are believed to negatively influence a wide range of mechanical and physiological parameters such as muscle strength, range of motion, and symmetry, what could potentially influence sports performance.

Spinal Manipulative Therapy (SMT) is a safe and effective therapy for musculoskeletal disorders that has been increasingly utilized in sports. SMT purpose is to correct spinal joints biomechanical dysfunctions using a high-velocity, low-amplitude movement, applied at the paraphysiological space, beyond the passive joint range of motion.

Kinetic and kinematic symmetry can be measured in commonly utilized physical functional tests often used as indicators of athlete's performance. Symmetry Index calculation is used to verify bilateral asymmetries in static and dynamic tests.

DETAILED DESCRIPTION:
Therefore, the objective of this randomized controlled trial study is to measure the immediate effects of lumbar SMT on kinetic and kinematic symmetry of asymptomatic athletes, through of the use of three commonly used functional tests: Static posture, Free Squat, and Countermovement Jump (CMJ) are often used as indicators of athlete's performance. These quantitative data is important to assess training effectiveness and prevention/ rehabilitation programs outcomes. To our knowledge this is the first study on literature that measured the immediate effects of SMT on kinetic and kinematic symmetry.

ELIGIBILITY:
Inclusion criteria

The inclusion criteria for sample followed the assumptions below:

* All young student participants had to be of both sexes, age between 18-35 years old.
* All participants had to be pain free or asymptomatic, with regards to low back pain, in order to create homogeneity within the study sample.
* All participants had to have at least a minimal score, (low level) of physical activity, evaluated by (IPAQ) questionnaire (International Physical Activity Questionnaire). This was done on the argument that the minimal score, already shows that the participants were minimally physically active. This also contributed in an indirect way to assure a certain degree of sample homogeneity, scoring the minimal level of physical activity to include in the study;
* All participants were required to show the subluxations or vertebral dysfunctions in their lumbar spine, detected by motion palpation. Through the purposive sampling, was allowed participants to officially take part in the study.

Exclusion Criteria:

The exclusion criteria for sample followed the assumptions below:

* Participants who received medical, surgical or in addition manual interventions prior or during the study, were immediately excluded.
* Participants who presented with any contraindications to manipulation on spine, which included but was not limited to osteomyelitis, tuberculosis, infectious arthritis, disc extrusion, hemangioma, vertebral malignancy and advanced spondylolisthesis
* Participants who have participating of sports competitions or change in training routine during the collecting data, was immediately withdraw from the study.;
* Participants with no vertebral dysfunction in the palpated lumbar joints were excluded of the study;
* Participants who did not sign the informed consent form, or not agree of the conditions, or did not have conditions to compromise with the schedule, were immediately withdraw from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Kinetic Symmetry (Lower Limbs Ground Reaction Forces) | 5 min after lumbar SMT intervention
  Lower Limbs Ground Reaction Forces measured by the force platforms

SECONDARY OUTCOMES:
Kinematic Symmetry (Linear Global Joint Centers Vectors Displacement) | 5 min after lumbar SMT intervention
  Linear Global Joint Centers Vectors Displacement measured by the 3D motion capture system

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Alvarenga, Phd, Principal Investigator — ULisboa
Locations (1):
- Bruno Araújo Procópio de Alvarenga, Lisbon, Portugal

REFERENCES:
- [Derived] Alvarenga BAP, Fujikawa R, Joao F, Lara JPR, Veloso AP. The effects of a single session of lumbar spinal manipulative therapy in terms of physical performance test symmetry in asymptomatic athletes: a single-blinded, randomised controlled study. BMJ Open Sport Exerc Med. 2018 Nov 28;4(1):e000389. doi: 10.1136/bmjsem-2018-000389. eCollection 2018. PMID 30555714
- See also: The Biomechanics and Functional Morphology Laboratory (BFML) is a research and education facility within the Faculty of Human Kinetics (FMH) and the University of Lisbon (ULisboa). — http://neuromechanics.fmh.ulisboa.pt